CLINICAL TRIAL: NCT03149016
Title: Evaluation of Treatment Outcomes of Corticotomy-accelerated Upper Incisors' Retraction: A Randomized Controlled Trial
Brief Title: The Use of Corticotomy for Upper Incisors Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-02-2017
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticotomy-assisted Retraction (Experimental): Corticotomy-assisted retraction will be performed in order to help in accelerating upper incisors' retraction
  Interventions: Procedure: Corticotomy-assisted Retraction
- Conventional Retraction (No Intervention): Conventional retraction will be used in this group of patients by sliding mechanisms

INTERVENTIONS:
Procedure: Corticotomy-assisted Retraction — Using a tunneling technique, the researcher will perform the intervention in the alveolar bone surrounding the upper incisors before retraction.
  Arms: Corticotomy-assisted Retraction

SUMMARY:
We aim to assess the treatment outcomes following upper incisors retraction accelerated by corticotomy procedure. So, we intend to randomize orthodontic patients with class II division I malocclusion into two groups: experimental group and control group. Both groups will start orthodontic treatment. Once a 0.019*0.025-inch stainless steel wire is fully engaged to the brackets, 1st premolars will be extracted. Canines will be retracted in the conventional manner. Then, the actual evaluation period starts when the upper incisors are retracted using two different methods.

DETAILED DESCRIPTION:
In the last three decades, the number of adult patients seeking short orthodontic treatment time has apparently increased as the conventional orthodontic treatment usually lasts for 20-24 months. Furthermore, orthodontic treatment is often associated with root resorption, bone degradation and caries development. Patients nowadays desire to end the orthodontic treatment as soon as possible due to phsycosocial reasons and to get the goals of the treatment without affecting their social life .

So many tooth movement accelerating methods have been proposed. However, the surgical approached are considered the most effective and promising methods in accelerating tooth movement. The current research aims to evaluate the efficacy of the a new proposed surgical method compared to the conventional method in upper incisors' retraction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 15 to 27 years , with permanent dentition , without hypodontia .
* Overjet less than 10 mm
* Normal or increased growth pattern (Diagnosed by Y-axis angle)
* Mild to moderate crowding (Less than 3 mm)
* After canines retraction , at least 3 mm space should be available distal the lateral incisors
* Midline deviation shouldn't be more than 3 mm

Exclusion Criteria:

* Medically contraindicated patients to oral surgery .
* Existence of general health issue that affect orthodontic teeth movement
* Previous orthodontic treatment
* Mixed dentition
* Hypodontia (Except third molars)
* Bad oral hygiene

Ages: 15 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-20 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Rate of retraction | This will be measured at the completion of the retraction procedure, and is expected to take 2 months in the experimental group and four months in the control group.
  The distance that the incisors moved during retraction divided by the time required to retract the four upper incisors to their ideal positions.
Time required for retraction | This will be measured at the completion of the retraction procedure, and is expected to be within 2 months in the accelerated group and 4 months in the control group.
  The time required from the beginning of incisors' retraction till the the completion of this procedure.

SECONDARY OUTCOMES:
Change in the axial inclination of upper incisors | A radiograph will be taken at T1: one day before upper incisors' retraction and T2: one day after the completion of upper incisors' retraction. Completion of upper incisors' retraction is expected to be within 2 months in the accelerated group and 4 mo
  the angle between the long axis of the upper incisor and a reference plane drawn on a later cephalometric radiograph teken at two assessment times.
Anchorage loss | This will be measured one day following the completion of retraction of the upper four incisors using plaster study models and is expected to be within 2 months in the accelerated group and 4 months in the control group
  the amount of anchorage loss (in mm), which is the distance from a perpendicular line to the midpalatal suture and extends between central fossa of both upper first molars to the third palatal rugae . These measurements are made on plaster study models.
Root resorption | An panoramic image will be taken at T1: one day before the commencement of incisor retraction and T2: one day following the completion of retraction and is expected to be within 2 months in the accelerated group and 4 months in the control group
  This variable is related to the amount of incisor root resorption after treatment in both groups. This is measured on a panoramic image. The amount of root resorption = the length of an incisor after retraction subtracted from the length of an incisor before retraction. Two radiogrpahs are needed.

CONTACTS AND LOCATIONS:
Overall Officials: Ghaith Al Imam, DDS, Principal Investigator — MSc student in Orthodontics, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aboul-Ela SM, El-Beialy AR, El-Sayed KM, Selim EM, El-Mangoury NH, Mostafa YA. Miniscrew implant-supported maxillary canine retraction with and without corticotomy-facilitated orthodontics. Am J Orthod Dentofacial Orthop. 2011 Feb;139(2):252-9. doi: 10.1016/j.ajodo.2009.04.028. PMID 21300255
- [Background] Al-Naoum F, Hajeer MY, Al-Jundi A. Does alveolar corticotomy accelerate orthodontic tooth movement when retracting upper canines? A split-mouth design randomized controlled trial. J Oral Maxillofac Surg. 2014 Oct;72(10):1880-9. doi: 10.1016/j.joms.2014.05.003. Epub 2014 May 14. PMID 25128922
- [Background] Choo H, Heo HA, Yoon HJ, Chung KR, Kim SH. Treatment outcome analysis of speedy surgical orthodontics for adults with maxillary protrusion. Am J Orthod Dentofacial Orthop. 2011 Dec;140(6):e251-62. doi: 10.1016/j.ajodo.2011.06.029. PMID 22133959
- [Background] Chung KR, Kim SH, Lee BS. Speedy surgical-orthodontic treatment with temporary anchorage devices as an alternative to orthognathic surgery. Am J Orthod Dentofacial Orthop. 2009 Jun;135(6):787-98. doi: 10.1016/j.ajodo.2007.03.036. PMID 19524840
- [Background] Bhattacharya P, Bhattacharya H, Anjum A, Bhandari R, Agarwal DK, Gupta A, Ansar J. Assessment of Corticotomy Facilitated Tooth Movement and Changes in Alveolar Bone Thickness - A CT Scan Study. J Clin Diagn Res. 2014 Oct;8(10):ZC26-30. doi: 10.7860/JCDR/2014/9448.4954. Epub 2014 Oct 20. PMID 25478442
- [Background] Dincer M, Gulsen A, Turk T. The retraction of upper incisors with the PG retraction system. Eur J Orthod. 2000 Feb;22(1):33-41. doi: 10.1093/ejo/22.1.33. PMID 10721243
- [Background] KOLE H. Surgical operations on the alveolar ridge to correct occlusal abnormalities. Oral Surg Oral Med Oral Pathol. 1959 May;12(5):515-29 concl. doi: 10.1016/0030-4220(59)90153-7. No abstract available. PMID 13644913